CLINICAL TRIAL: NCT02016872
Title: Prognostic Value of Tumor Hypoxia, as Measured by 18F-FMISO Breath Hold PET/CT, in Non-Small-Cell-Lung Cancer (NSCLC) Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 13-186; U01CA157442-01A1 (NIH)
Record Dates: First submitted 2013-12-16; First posted 2013-12-20 (Estimated); Results first posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2024-07

CONDITIONS: Non-Small-Cell-Lung Cancer (NSCLC)
Keywords: PET/CT; 18F-FMISO; tumor hypoxia; 13-186
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — fluoromisonidazole

ARMS (1):
- 18F-FMISO PET/CT (Experimental): All enrolled patients will undergo a baseline 18F-FDG PET scan as part of their standard clinical treatment for NSCLC. Dynamic 18F-FMISO PET scans will be performed on one of the GE PET/CT scanners in 3D mode, at least one day after the baseline 18F-FDG PET scan. The dynamic baseline 18F-FMISO studies may precede the 18F-FDG study if the patient had a CT or PET/CT scan within the last 30 days that would permit the investigators to localize the tumor of interest during the 18F-FMISO study. In a group of 5 patients, the feasibility of simultaneous imaging of 18F-FMISO and 18F-FDG will be assessed. The patient will have an IV line placed for radiotracer injection and for venous blood sampling. All dynamic PET scans will be performed over one PET FOV centered at the lesion position. The 18F-FDG mid-treatment PET/CT scan will be performed over only one bed position.
  Interventions: Drug: 18F-FMISO; Other: PET/CT

INTERVENTIONS:
Drug: 18F-FMISO
Other: PET/CT

SUMMARY:
The purpose of this study is to help researchers investigate if a new imaging agent named 18F-FMISO can predict if patients with lung cancer will respond to standard therapy, as well as whether disease will reoccur in the future. The study will also investigate whether a 18F-FDG PET scan in the middle of radiation treatment can predict if lung cancer will respond to standard therapy. Information obtained from this study may help doctors design future studies in which they may target tumor areas that do not respond to therapy or may likely reoccur in the future.

ELIGIBILITY:
Inclusion Criteria:

* Pathologic confirmation of NSCLC at MSKCC
* No prior treatment for this diagnosis of NSCLC
* Patient to be treated with neoadjuvant chemotherapy (35 patients total) or patient to be treated with definitive RT,sequential chemo-RT, or concurrent chemo-RT (minimum dose of 50 Gy in 25 fractions) (25 patients total)
* Tumor must measure ≥ 2cm on CT
* Age ≥ 18 years
* Ability to hold the breath for 10 seconds.
* Karnofsky performance status ≥ 70%
* Women of childbearing age must have a negative blood pregnancy test

Exclusion Criteria:

* Women who are pregnant or breast-feeding
* Severe diabetes (fasting Blood Glucose > 200 mg/dl)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2013-12-16 (Actual); Primary Completion 2024-07-08 (Actual); Study Completion 2024-07-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Shin, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Derived] Grkovski M, Schwartz J, Rimner A, Schoder H, Carlin SD, Zanzonico PB, Humm JL, Nehmeh SA. Reproducibility of 18F-fluoromisonidazole intratumour distribution in non-small cell lung cancer. EJNMMI Res. 2016 Dec;6(1):79. doi: 10.1186/s13550-016-0210-y. Epub 2016 Nov 7. PMID 27822900
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- 18F-FMISO PET/CT: All enrolled patients will undergo a baseline 18F-FDG PET scan as part of their standard clinical treatment for NSCLC. Dynamic 18F-FMISO PET scans will be performed on one of the GE PET/CT scanners in 3D mode, at least one day after the baseline 18F-FDG PET scan.
Period: Overall Study
Arm/Group | 18F-FMISO PET/CT
Started | 25
Completed | 10
Not Completed | 15
Not completed — Withdrawal by Subject | 10
Not completed — Death Progression | 2
Not completed — No FMISO scan | 1
Not completed — Ineligible | 2

BASELINE CHARACTERISTICS:
Arm/Group | 18F-FMISO PET/CT
Number analyzed (Participants) | 25
Age, Continuous [Mean (Full Range); unit: years] | 64 [30 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 22
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 17
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: The Difference Between Two Baseline Fluorine-18-labeled Fluoro-misonidazole (18F-FMISO) Scans
Description: The difference between two baseline 18F-FMISO PET scans three days apart to assess the reproducibility.
Time Frame: 3 days from baseline
Population: Participants who completed study treatment
Measure: Number (95% Confidence Interval); unit: unitless
Arm/Group | 18F-FMISO PET/CT
Number analyzed (Participants) | 10
unitless
  k1 | 0 [-0.1190 to 0.1203]
  k3 | 0 [-0.0159 to 0.0146]

2. Primary Outcome: Progression-free Survival (PFS)
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: 3 years
Population: Participants who completed study treatment
Measure: Number; unit: % of pts with progression free survival
Arm/Group | 18F-FMISO PET/CT
Number analyzed (Participants) | 10
% of pts with progression free survival | 58.3

3. Secondary Outcome: Overall Survival
Time Frame: 3 years
Population: Participants who completed study treatment
Measure: Number; unit: % of participants alive
Arm/Group | 18F-FMISO PET/CT
Number analyzed (Participants) | 10
% of participants alive | 40

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | 18F-FMISO PET/CT
All-Cause Mortality (participants affected / at risk) | 6/25
Serious Adverse Events (participants affected / at risk) | 2/25
Other Adverse Events (participants affected / at risk) | 2/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 18F-FMISO PET/CT (N=25)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Non-cardiac chest pain secondary to migration of esophageal stent (General disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 18F-FMISO PET/CT (N=25)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Non-cardiac chest pain secondary to migration of esophageal stent (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-12-22): https://cdn.clinicaltrials.gov/large-docs/72/NCT02016872/Prot_SAP_000.pdf